CLINICAL TRIAL: NCT05944679
Title: Prospective Randomized Study of the Clinical Utility to Follow-up Radiographs During the First Year of Knee Replacement Surgery
Brief Title: Clinical Utility to Follow-up Radiographs During the First Year of Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Pelfort Lopez, Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Radioprotesi
Record Dates: First submitted 2023-06-27; First posted 2023-07-13 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Prosthetic Knee Surgery
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Xray (Placebo Comparator): Xray at 1, 3, 6 and 12 months
  Interventions: Radiation: Xray
- Group No Xray (Active Comparator): Xray at 12 months
  Interventions: Radiation: No Xray

INTERVENTIONS:
Radiation: No Xray — Just one Xray 12 months after the intervention
  Arms: Group No Xray
Radiation: Xray — Xray at 1, 3, 6 and 12 months after intervention
  Arms: Group Xray

SUMMARY:
Primary prosthetic surgery for the treatment of gonarthrosis is currently one of the most prevalent surgical treatments in Traumatology. The Arthroplasty Register in Catalonia, which started in 2005, counted more than 60.000 knee prothesis until 2015. Regarding the peridiocity for taking control radiographs in patients undergoing knee replacement surgery, there is no consensus. This means, that in similar studies that evaluate the results of prosthetic surgery, there is a great variability in radiological follow-up protocols, especifically during the firts post-operative years. Given the high prevalence and the long survival period demonstrated by these implants, it seems reasonable to be able to establish the real value of the radiographs performed during the first year of follow-up after surgery. From this perspective, the aim of our study is to evaluate if conducting just two radiographs instead of five during the first postoperative year after the surgery, has any influence on the clinical and functional results of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily agree to be part of the study and sign the informed consent
* Patients awaiting prosthetic knee surgery with a diagnosis of gonarthrosis without age limit (>18 years)
* All cases of prothesis cemented to the tibia and femur will be included, regardless of whether or not the patellar component is prosthetic
* Patients with knee prothesis and cruciate ligament retention, with ultracongruent polyethylene or posterostabilized as a maximum degree of prosthetic constriction
* The implants will be the usual ones used in our Center for primary prosthetic knee surgery, Journey (smith-Nephew) and Persona or NexGen (Zimmer)

Exclusion Criteria:

* Patients who do not voluntariily agree to participate
* Patients undergoing primary prosthetic surgery in relation to tibial plate fractures
* Patients awaiting a unicompartimental or patellofemoral prothesis
* Patients who, for any reason, want to leave the study during the follow-up period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
KSS Test change | Preoperative, 6 and 12 months
  Change value from preoperative condition to 12 months after operation, including 6 month assessment
KOOS Test change | Preoperative, 6 and 12 months
  Change value from preoperative condition to 12 months after operation, including 6 month assessment
SF-12 Test change | Preoperative, 6 and 12 months
  Change value from preoperative condition to 12 months after operation, including 6 month assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans JT, Walker RW, Evans JP, Blom AW, Sayers A, Whitehouse MR. How long does a knee replacement last? A systematic review and meta-analysis of case series and national registry reports with more than 15 years of follow-up. Lancet. 2019 Feb 16;393(10172):655-663. doi: 10.1016/S0140-6736(18)32531-5. Epub 2019 Feb 14. PMID 30782341
- [Background] Gomez-Valero S, Garcia-Perez F, Florez-Garcia MT, Miangolarra-Page JC. A systematic review of self-administered questionnaires for the functional assessment of patients with knee disabilities adapted into Spanish. Rev Esp Cir Ortop Traumatol. 2017 Mar-Apr;61(2):96-103. doi: 10.1016/j.recot.2016.11.002. Epub 2017 Jan 31. English, Spanish. PMID 28159566
- [Background] Walker LC, Clement ND, Bardgett M, Weir D, Holland J, Gerrand C, Deehan DJ. The WOMAC score can be reliably used to classify patient satisfaction after total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2018 Nov;26(11):3333-3341. doi: 10.1007/s00167-018-4879-5. Epub 2018 Feb 26. PMID 29484445
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Meneghini RM, Mont MA, Backstein DB, Bourne RB, Dennis DA, Scuderi GR. Development of a Modern Knee Society Radiographic Evaluation System and Methodology for Total Knee Arthroplasty. J Arthroplasty. 2015 Dec;30(12):2311-4. doi: 10.1016/j.arth.2015.05.049. Epub 2015 May 29. PMID 26122112
- [Background] Rissolio L, Sabatini L, Risitano S, Bistolfi A, Galluzzo U, Masse A, Indelli PF. Is It the Surgeon, the Patient, or the Device? A Comprehensive Clinical and Radiological Evaluation of Factors Influencing Patient Satisfaction in 648 Total Knee Arthroplasties. J Clin Med. 2021 Jun 12;10(12):2599. doi: 10.3390/jcm10122599. PMID 34204628
- [Background] Sarmah SS, Patel S, Hossain FS, Haddad FS. The radiological assessment of total and unicompartmental knee replacements. J Bone Joint Surg Br. 2012 Oct;94(10):1321-9. doi: 10.1302/0301-620X.94B10.29411. PMID 23015555
- [Background] Ewald FC. The Knee Society total knee arthroplasty roentgenographic evaluation and scoring system. Clin Orthop Relat Res. 1989 Nov;(248):9-12. PMID 2805502
- [Background] Khalifa AA, Mullaji AB, Mostafa AM, Farouk OA. A Protocol to Systematic Radiographic Assessment of Primary Total Knee Arthroplasty. Orthop Res Rev. 2021 Jul 17;13:95-106. doi: 10.2147/ORR.S320372. eCollection 2021. PMID 34305412
- [Background] Baek JH, Lee SC, Choi K, Ahn HS, Nam CH. Long-term survivorship of total knee arthroplasty with a single-radius, high-flexion posterior stabilized prosthesis. Knee. 2021 Jun;30:275-282. doi: 10.1016/j.knee.2021.04.017. Epub 2021 May 11. PMID 33984746
- [Background] Miralles-Munoz FA, Rubio-Morales M, Bello-Tejada L, Gonzalez-Parreno S, Lizaur-Utrilla A, Alonso-Montero C. Varus alignment of the tibial component up to seven degrees is not associated with poor long-term outcomes in a neutrally aligned total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2022 Aug;30(8):2768-2775. doi: 10.1007/s00167-021-06627-3. Epub 2021 Jun 26. PMID 34175990
- [Background] Sabatini L, Aprato A, Camazzola D, Bistolfi A, Capella M, Masse A. Primary total knee arthroplasty in tibial plateau fractures: Literature review and our institutional experience. Injury. 2023 Mar;54 Suppl 1:S15-S23. doi: 10.1016/j.injury.2021.02.006. Epub 2021 Feb 7. PMID 33583591
- [Background] Webb JI, Stoner RS, Afzal I, Evans CR, Scott G, Field RE. The Medial Rotation Knee replacement: Clinical and radiological results of a multi-centre surveillance study at five years. Knee. 2021 Jan;28:247-255. doi: 10.1016/j.knee.2020.12.025. Epub 2021 Jan 13. PMID 33453513
- [Background] Glaser D, Lotke P. Cost-effectiveness of immediate postoperative radiographs after uncomplicated total knee arthroplasty: a retrospective and prospective study of 750 patients. J Arthroplasty. 2000 Jun;15(4):475-8. doi: 10.1054/arth.2000.4338. PMID 10884208
- [Background] Hassan S, Wall A, Ayyaswamy B, Rogers S, Mills SP, Charalambous CP. Is there a need for early post-operative x-rays in primary total knee replacements? Experience of a centre in the UK. Ann R Coll Surg Engl. 2012 Apr;94(3):199-200. doi: 10.1308/003588412X13171221501780. PMID 22507727
- [Background] Novack TA, Patel JN, Koss J, Mazzei C, Harrington CJ, Wittig JC, Dundon J. Is There a Need for Recovery Room Radiographs Following Uncomplicated Primary Total Knee Arthroplasty? Cureus. 2021 Apr 18;13(4):e14544. doi: 10.7759/cureus.14544. PMID 34017659
- [Background] Aljawder A, Alomran D, Alayyoub M, Alkhalifa F. Immediate Postoperative Portable Radiograph After Total Knee Replacements: A Necessity or a Burden? Open Orthop J. 2018 May 31;12:173-179. doi: 10.2174/1874325001812010173. eCollection 2018. PMID 29997704